CLINICAL TRIAL: NCT05695677
Title: Capacitive-Resistive Radiofrequency Therapy of the Neck Muscles as a Non-invasive Treatment of the Post-dural Puncture Headache After Cesarean Delivery. A Pre-post Study.
Brief Title: Radiofrequency Therapy of the Neck Muscles for Treating the Post-dural Puncture Headache After Cesarean Delivery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MS-254-2022
Record Dates: First submitted 2022-10-18; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Tecar Therapy Efficacy in the Treatment of PDPH

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tecar treatment sucess (Other)
  Interventions: Procedure: Capacitive-Resistive Radiofrequency therapy of the neck muscles

INTERVENTIONS:
Procedure: Capacitive-Resistive Radiofrequency therapy of the neck muscles — Capacitive-Resistive Radiofrequency therapy of the neck muscles as a non-invasive technique for treating PDPH.

SUMMARY:
Postdural puncture headache (PDPH) is a frequent complication after neuraxial anaesthesia due to accidental puncture of the dura mater. After spinal anaesthesia, the rate of PDPH may reach up to 28,7% of cases. PDPH is more common in females, especially obstetric patients, young age and more after epidural than spinal anaesthesia because of needle type. PDPH interferes with the patient's ability to resume activities, prolongs the hospital stay, and causes chronic headaches in up to 28% of cases.

Several treatment modalities were described for PDPH. Conservative treatment, an epidural blood patch, peripheral nerve blocks, such as sphenopalatine ganglion block (SPGB) and more excellent occipital nerve block (GONB) using local anaesthetic block or through percutaneous radiofrequency ablation or direct injection of local anaesthetic and steroid directly into the neck muscles; were all proven effective in treating PDPH. Radiofrequency (RF) is a commonly used technique to treat different types of pain, headaches, and musculoskeletal abnormalities. The second-generation non-invasive RF modality was recently developed as Tecar therapy (TECAR: Capacitive and Resistive Energy Transfer). Tecar therapy provided promising results in treating chronic pelvic and postpartum perineal pain. To our knowledge, Tecar therapy efficacy in treating PDPH has not been evaluated before. This study aims to assess the effectiveness of Tecar therapy as a non-invasive technique for treating PDPH. This study hypothesizes that Tecar therapy could be an effective non-invasive technique for treating or reducing PDPH.

ELIGIBILITY:
Inclusion Criteria:

* female patients aged over 18 years
* ASA physical status I or II.
* scheduled for elective cesarean delivery under spinal anaesthesia
* who developed PDPH with failed conservative treatment

Exclusion Criteria:

* Patients with a history of long-standing diabetes.
* peripheral vascular diseases
* cervical spine disorders
* receiving analgesics and anticonvulsant medication .

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
is the rate of Tecar therapy success in treating the PDPH after the first session | starting from day 2 after developing PDPH and over 5 days.
  number of patients with VAS <4 in sitting position after the first session / total number of patients).

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Ahmed, MD, Principal Investigator — kasr Alainy Faculty of medicine
Locations (2):
- Egypt (2):
  - Abeer Ahmed, Cairo
  - Anesthesia department - Faculty of medicine- Cairo University, Cairo